CLINICAL TRIAL: NCT02815618
Title: An Optical Neuro-monitor of Cerebral Oxygen Metabolism and Blood Flow for Neonatology
Acronym: BabyLux
Status: Completed | Type: Observational
Sponsor: Gorm Greisen (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, Professor, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: BabyLux CIP 4.1
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Hemodynamic Instability
Keywords: Time-resolved spectroscopy; Diffuse correlation spectroscopy; Neonatology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Infants delivered by elective caesarean: Infants to be measured immediately after birth and on their second day of life.
  Interventions: Device: BabyLux Neuro-monitor
- Infants on mechanical ventilation: Infants to be measured while changing ventilator settings to normalize arterial pCO2.
  Interventions: Device: BabyLux Neuro-monitor
- Infants on ventilatory support: Infants to be measured for 24 hours continuously to assess user-friendliness and loss of signal.
  Interventions: Device: BabyLux Neuro-monitor

INTERVENTIONS:
Device: BabyLux Neuro-monitor — Measurement of cerebral blood flow index (CBFi) and tissue oxygen saturation (StO2).

SUMMARY:
Feasibility trial on the use of a hybrid optical device integrating time-resolved near-infrared spectroscopy (TRS) and diffuse correlation spectroscopy (DCS) for measurement of cerebral oxygen metabolism and blood flow in neonates.

The device wil be tested in four settings measuring:

1. Changes in cerebral oxygenation and haemodynamics after birth
2. precision and repeatability
3. The cerebral vaso-reactivity to arterial carbon dioxide
4. Assessment of the user-friendliness and loss of signal in routine care

DETAILED DESCRIPTION:
The BabyLux project aims to provide a precise, accurate, and robust device to continuously monitor cerebral oxygen metabolism and blood flow in critically ill newborn infants. This will be achieved by combining time resolved near-infrared spectroscopy (TRS) with newly developed diffuse correlation spectroscopy (DCS) in a single device. The innovative aspects of the project are related to the use of advanced solutions, based on state-of-the-art photonic components, which have already been tested in laboratory and clinical tests on adults.

Time Resolved Near-infrared spectroscopy and Diffuse Correlation Spectroscopy

The proposed solution will integrate two advanced photonic techniques, TRS and DCS. Both techniques rely on the use of an optical fibre probe (sensor) to illuminate with very low power near-infrared light the scalp and to collect the diffusively reflected optical signal that has propagated through the scalp and skull, and therefore carries information on the deeper cortical region. The different absorption spectra of oxygenated and deoxygenated haemoglobin in the near-infrared range allows for the non-invasive monitoring of the two species in the cortical tissue.

TRS and DCS prototypes are available and have been technically tested in laboratory settings and successfully validated during preclinical trials on adult volunteers and patients.

Measured TRS/DCS parameters

TRS measures the attenuation and the temporal broadening of relatively short light pulses (pulse duration ~100 ps) through a diffusive medium (e.g. a neonate's head). TRS has the ability to resolve path-lengths (or equivalently time-of-flights) of photons that have propagated through the tissues. This enables TRS to separate the absorption and scattering coefficients allowing for absolute measurements, and to utilize time-gating of path-lengths to emphasize signals from deeper tissues. This is particularly important for separating intra- and extra-cerebral signals for brain monitoring.

DCS relies on the fact that temporal correlation of light fields in turbid media also obeys a diffusion equation, albeit a slightly different one than is used for TRS. Thus DCS shares the light penetration advantages of TRS, but, since DCS explicitly measures red blood cell movement, it provides a direct measure of quantities such as cerebral blood flow (CBF).

The specific combination of DCS and TRS allows for the assessment of cerebral oxygen metabolism and CBF in a complete (i.e. CBF and oxygenation are simultaneously and independently provided), accurate (i.e. based on absolute measurements of optical parameters) and robust (i.e. potentially less affected by artefacts related to superficial systemic activity or sensor/head movements) way.

The aim of this study is to perform clinical measurements using the BabyLux instrument in different clinical real-life settings to validate this new technology in terms of feasibility, repeatability of measurements, and user friendliness in neonatal medicine.

The BabyLux system is tested in four different real-life settings to measure:

1. The increase in oxygenation and change in blood flow during the minutes after birth to specify the expected range of measurement;
2. The precision and repeatability of measurements by reapplying the NIRS sensor several times on slightly different sites of the head in a relatively steady condition;
3. The cerebral vaso-reactivity to arterial carbon dioxide tension in mechanically ventilated newborns to monitor induced changes in cerebral blood flow;
4. The user-friendliness and loss of signal in routine care situations (e.g. during 24-hour monitoring of neonates undergoing intensive care).

ELIGIBILITY:
Setting 1 and 2:

Inclusion Criteria:

* GA > 37 weeks
* planned to be delivered by an uncomplicated elective caesarean section

Exclusion Criteria:

* need for resuscitation or supplementary oxygen during the first 10 minutes following umbilical cord clamping
* congenital malformations

Setting 3:

Inclusion Criteria:

* GA < 37 weeks
* Postnatal age more > 24 hours
* Mechanically ventilated
* Clinically stable
* Normal brain ultrasound
* Transcutaneous pCO2 monitoring (tcpCO2)

Exclusion Criteria:

* Congenital malformations

Setting 4:

Inclusion Criteria:

* Postnatal age < 28 days
* ventilatory support by mechanical ventilation or nasal CPAP

Exclusion Criteria:

* Congenital malformations

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Setting 1 and 2:
  Newborn infants immediately after delivery by elective caesarean and on their second day of life.
  Setting 3:
  Premature infants on mechanical ventilation.
  Setting 4:
  Neonate infants on ventilatory support
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation (StO2) after birth. | 10 min immediately after umbilical cord clamping.
  Measurement of cerebral haemodynamics immediately after birth.
Precision and repeatability | During second day of life.
  Test-retest variability estimated by within-subject standard deviation in one-way ANOVA with subject as factor.
Cerebral vaso-reactivity to arterial carbon dioxide | 1 hour after change in ventilator settings.
  Mean CBFi and tcpCO2 one minute before the change and 15 min after will be used to analyse CBFi-tcpCO2 reactivity.
Assessment of user-friendliness and loss of signal in routine care | 24 hours of contineous measurements.
  Assessed by Likert-scale questionnaire completed by clinical staff.

CONTACTS AND LOCATIONS:
Overall Officials: Gorm Greisen, MD, Prof., Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Carli A, Andresen B, Giovannella M, Durduran T, Contini D, Spinelli L, Weigel UM, Passera S, Pesenti N, Mosca F, Torricelli A, Fumagalli M, Greisen G. Cerebral oxygenation and blood flow in term infants during postnatal transition: BabyLux project. Arch Dis Child Fetal Neonatal Ed. 2019 Nov;104(6):F648-F653. doi: 10.1136/archdischild-2018-316400. Epub 2019 May 13. PMID 31085677
- See also: The BabyLux project web-site — http://www.babylux-project.eu